CLINICAL TRIAL: NCT00162292
Title: Multiple Ascending Dose Study of BMS-582949 in Patients With Stable Rheumatoid Arthritis on the Methotrexate Background
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Study Director, Bristol-Myers Squibb
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IM119-010
Record Dates: First submitted 2005-09-09; First posted 2005-09-13 (Estimated); Last update posted 2010-03-02 (Estimated); Status verified 2008-08

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — 4-(5-(cyclopropylcarbamoyl)-2-methylphenylamino)-5-methyl-N-propylpyrrolo(1,2-f)(1,2,4)triazine-6-carboxamide; Methotrexate

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Drug: BMS-582949 and Methotrexate

SUMMARY:
The purpose of this clinical research study is to learn if it is safe for rheumatoid arthritis patients to take BMS-582949 along with methotrexate.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-70 years
* Diagnosis of RA for ≥6 months
* Swollen or tender joint or ESR >ULN. Subject must be on stable doses of MTX
* Women of Childbearing Potential

Exclusion Criteria:

* Serum transaminase levels >ULN
* CK>ULN
* Cannot have taken Orencia or Remicade within 8 weeks of baseline, Humira or Enbrel within 4 weeks of baseline
* Use of H2 blockers or Proton Pump inhibitors while on study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Estimated)
Dates: Start 2005-11; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
To evaluate safety and tolerability of BMS-582949 in subjects with active rheumatoid arthritis receiving concomitant MTX at steady state | during 28 doses of treatment

SECONDARY OUTCOMES:
To evaluate the PK of BMS-582949 in clinically stable RA subjects on stable doses of MTX and concomitant BMS-582949
To explore DAS28, ESR, RF and CRP of clinically stable doses of MTX and concomitant BMS-582949 compared to MTX alone | during 28 days of treatment
To evaluate PK of MTX in stable RA subjects in the absence and presence of BMS-582949 for subjects enrolled prior to approval of amendment 2

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (10):
- United States (8):
  - Desert Medical Advances, Palm Desert, California
  - Boling Clinical Trials, Upland, California
  - Delray Research Associates, Delray Beach, Florida
  - Ocala Rheumatology Research Center, Ocala, Florida
  - Phase Iii Clinical Research, Fall River, Massachusetts
  - Covance Clinical Research Unit Inc., Dallas, Texas
  - Radiant Research San Antonio Northeast, San Antonio, Texas
  - Healthcare Discoveries, Inc, San Antonio, Texas
- Mexico (2):
  - Local Institution, León, Guanajuato
  - Local Institution, Metepec, State of Mexico